CLINICAL TRIAL: NCT06733987
Title: Immunological Senescence Phenotype as a Resistance Profile to Pembrolizumab in Patients With Relapsed/Refractory Hodgkin's Lymphoma
Acronym: HL-SIP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: HL-SIP; funding number not available (Other Grant/Funding Number: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2024-12-01; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hodgkin Lymphoma
Keywords: pembrolizumab
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The haematological and haematochemical examinations required by clinical practice for patients included in the study will be performed. Study-specific blood samples will be taken at the same time as the clinical practice samples.
  Cytofluorimetric and molecular investigations will be performed at the Laboratory of Transplantation Immunobiology and Advanced Cellular Therapies (IBT) of the IRCCS AOU of Bologna.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-centre, observational, prospective and exploratory study, which involves the use of human tissues from patients affected by Relapsed/Refractory classic Hodgkin Lymphoma treated with pembrolizumab at the Departmental Diagnosis and Therapy program for chronic lymphoproliferative syndromes of the IRCCS AOU of Bologna. Peripheral blood samples will be used for the study and will be taken:

* before starting treatment with pembrolizumab.
* undergoing therapy with pembrolizumab (cycle 2 (C2), C3, C4, C8, C12).

DETAILED DESCRIPTION:
This is a single-centre, observational, prospective and exploratory study using human tissues from cHL R/R patients treated with pembrolizumab at the IRCCS AOU of Bologna's Diagnosis and Therapy of Chronic Lymphoproliferative Syndromes Departmental Programme. Peripheral blood samples will be used for the study

* before starting treatment with pembrolizumab.
* during pembrolizumab therapy (cycle 2 (C2), C3, C4, C8, C12). Patients who have achieved complete metabolic remission will continue pembrolizumab for two years without any consolidation therapy, while those who have achieved a partial response (after about 14-16 doses) will receive allo-transplantation.

Withdrawals will be performed according to clinical practice in accordance with the doctor's judgement. The diagnostic-therapeutic course of the patients will in no way be influenced by the outcome of the tissue examinations that will be carried out for the purposes of the study.

All patients with cHL R/R who are candidates for treatment with pembrolizumab as part of the normal care pathway at the IRCCS AOU of Bologna's Diagnosis and Treatment of Chronic Lymphoproliferative Syndromes Departmental Programme will be prospectively enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged ≥ 18 years at enrollment
* Patients affected by cHL R/R candidate to receive a treatment with Pembrolizumab
* Signature of informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population includes (R/R) cHL patients who receive a treatment with Pembrolizumab at the Unit of Hematology, IRCCS-Azienda Ospedaliero-Universitaria of Bologna
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
correlation between immunological profile of SIP and response to pembrolizumab | At the end of Cycle 2 (each cycle is 21 days)
  Cytofluorimetric characterisation

SECONDARY OUTCOMES:
The correlation of cfDNA with response to therapy | during pembrolizumab therapy (cycle 2, 3, 4, 8 and12, each cycle is 21 days), through study completion, an average of 2 year
  Clinical response: absence of clinical signs and symptoms of disease according to international criteria (Cheson et al 2007) and assessed by PET/CT examination. Metabolic response: negative uptake in PET/CT or Deauville scale <3
The correlation of peculiar mutations with response to therapy | during pembrolizumab therapy (cycle 2, 3, 4, 8 and12, each cycle is 21 days), through study completion, an average of 2 year
  Clinical response: absence of clinical signs and symptoms of disease according to international criteria (Cheson et al 2007) and assessed by PET/CT examination. Metabolic response: negative uptake in PET/CT or Deauville scale <3

CONTACTS AND LOCATIONS:
Overall Officials: Pier Luigi Zinzani, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No